CLINICAL TRIAL: NCT04787185
Title: STRAIT-LUC Trial: Stereotactic Radiotherapy (SRT) in Association With Immunotherapy for the Treatment of Brain Metastases From Non-small Cell Lung Cancer (NSCLC): a Multicenter Prospective Observational Study
Brief Title: Stereotactic Radiotherapy in Association With Immunotherapy for the Treatment of NSCLC Brain Metastases
Acronym: STRAITLUC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Lorenzo Livi, Professor, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 15901
Record Dates: First submitted 2020-12-22; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Brain Metastases From NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Valutation of toxicity — Observation of toxicity
  All patient with Brain metastases from NSCLC who are candidates for RS or HFSRT in course of immunotherapy

SUMMARY:
The study's primary objective is the evaluation of toxicities reported during RS or HFSRT in patients with brain metastases from NSCLC undergoing immunotherapy (Safety), with particular reference to the rate of symptomatic radionecrosis and intralesional hemorrhage. Others primary objectives of the study are the Feasibility and the intracranial control of the disease, both local (site radiotherapy treatment) and at a distance (intracranial, but at a distance from the site of the disease treated with stereotaxic radiotherapy). The secondary objectives concern quality assessment of life of the patients under study (Quality Of Life, QoL).

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years

  * Ability to express informed consent
* Histological or cytological diagnosis (possibility of PDL-1 determination) of NSCLC
* - Brain metastases up to a maximum of 10 and all treated with RS or Hypofractionated stereotactic radiotherapy (3 to 5 fractions)
* Brain disease assessable according to iRANO criteria
* Radiation therapy on brain metastases within 4 weeks before or after infusion of immunotherapy in the following settings
* brain metastases at initio brain metastases treated with RS + 1st line therapy
* Brain metastases as I progression after I line of systemic therapy CHT, IT or CHTIT regardless of whether or not the same line is continued (treatment Beyond progression) or shift to the next line;
* Brain metastases as II progression after II line of systemic therapy (CHT, IT) regardless of whether it is continued or not of the same line (treatment beyond progression) or shift to the next line.
* Diagnostic brain MRI for brain metastases within one month of treatment stereotactic

Esclusion criteria:

* Life expectancy of less than 6 months (calculated with GPA score <2)
* Performance Status> 2
* Previous radiotherapy treatment at the brain site
* Contraindication to MRI of the brain with contrast medium
* Presence of a number of intracranial metastases> 10
* Inability to express informed consent
* Infusion of immunotherapy more than 4 weeks before and after radiotherapy
* Impossibility of recording times and dosages of administration of steroid therapy
* Ineligibility for immunotherapy treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with brain metastasis for NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who experience grade 3-5 toxicity within 3 months of initiation, graded according to the National Cancer Institute (NCI) CTCAE version (v)4.0 | 24 Months
  Evaluation of toxicity related to the combination of radiotherapy and immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Radioterapia Oncologica AOU Careggi, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF